CLINICAL TRIAL: NCT04805294
Title: Coaching a Wellbeing Leadership Culture: Bringing a Pediatrician Wellbeing Program Into Practice
Brief Title: Pediatrician Wellbeing Program
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0987
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Burn Out; Burn Out (Psychology); Work Related Stress
Keywords: Wellbeing; Burn Out; Physician Burn Out; Mindfulness
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to implement a comprehensive Pediatrician Wellbeing Program initiated through and aligning with departmental faculty development and mentorship processes and goals. The Investigators hypothesize that a wellbeing intervention that incorporates an innovative health coaching model to cultivate individual behavior change supportive of one's own and others' wellbeing will lead to improvements in self-reported wellbeing.

DETAILED DESCRIPTION:
The investigators hypothesize that a wellbeing intervention that incorporates an innovative health coaching model to cultivate individual behavior change supportive of one's own and others' wellbeing can be implemented using existing institutional infrastructure and will lead to improvements in self-reported wellbeing.

This is a nonrandomized pilot study of a convenience sample. Participants will be assigned to 1 of 2 coaches, based upon availability of schedules. Participants who perform research will be assigned to the remote coach whenever possible to avoid potential concerns with the internal coach's dual role as Administrative Director of the Children's Research Institute.

The sample size for this pilot study (up to 30) was selected for feasibility and not power. This study is funded for 1-year and study participation is for 6-months. The study will be conducted at a single site; the University of North Carolina Department of Pediatrics Chapel Hill. Assistant, Associate and Full Professors, tenure-track or fixed-term, on the UNC main campus are eligible.

The Pediatric Wellbeing Program consists of coaching sessions from a certified National Board for Health and Wellness Coach (NBHWC) through the National Board of Medical Examiners. The NBHWC pioneered science-based training, education, and research of health and wellness coaches over the past 15 years. NBHWC became an accredited institution through National Board of Medical Examiners in 2016, providing certification through examination. By using NBHWC-certified coaches, the investigators are adhering to a standard and measured foundational competencies: the knowledge, tasks and skills essential to the practice of health and wellness coaching. Coaches will assist participants in constructing their Wellbeing-Individual Development Plan (Wellbeing-IDP). The Wellbeing-IDP is designed to assist with identifying the participant's vision, goals, and plan for wellbeing; assess current wellbeing with the WHO-5 to identify areas where they have high wellbeing and areas they need to develop; secure support and accountability (e.g., UNC resources, familial, peer, social, professional); and create a timeline for what they want to accomplish when.

As needed, faculty will also receive up to 5 additional coaching sessions from a certified health coach via video conferencing. All coaching sessions will use principles for health coaching, including brief motivational interviewing, self-empowerment and determination, transtheoretical model of stages of change, mindset, sense making, and making SMART goals (Specific, Measurable, Achievable, Relevant, Timely).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* An Assistant, Associate or Full Professor, either in fixed-term and tenure-track positions in the Department of Pediatrics on the UNC main campus, at the time of consent.

Exclusion Criteria:

* Not an Assistant, Associate or Full Professor in either fixed-term or tenure-track position within the Department of Pediatrics on the UNC main campus.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Assistant, Associate or Full Professor, either in fixed-term and tenure-track positions in the Department of Pediatrics on the UNC main campus, at the time of consent.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Persons Who Were Contacted to Enroll in the Study | through study completion, an average of 180 days
  Percentage of persons who were contacted to enroll in the study
Percentage of Persons Who Ultimately Enrolled in the Study | through study completion, an average of 180 days
  Potential persons who were contacted for study participation versus the number who ultimately enrolled in the study.
Percentage of Mentors Who Attended First Session | through study completion, an average of 180 days
  Percentage of mentors who attended first session with mentee
Percentage of Health Coach Visits Scheduled | through study completion, an average of 180 days
  Percentage of visits scheduled with health coaches
Percentage of Health Coach Visits Missed | through study completion, an average of 180 days
  Percentage of visits missed with health coaches
Percentage of Health Coach Visits Attended | through study completion, an average of 180 days
  Percentage of visits attended with health coaches
Percentage of Total Surveys Completed | Day 180
  Participants are asked to complete 6 surveys at baseline, 4 surveys after 3-months in the program and 7 surveys after 6-months in the program; the measure reports the number of fully executed surveys as a percentage to determine engagement.
Percentage of Participants Who Complete the Study | Day 180
  Percentage of participants who fully complete all visits and surveys in the study

SECONDARY OUTCOMES:
Change in World Health Organization Wellbeing Index (WHO-5) Scores | Day 1, Day 180
  The WHO-5 is a 5-item measure assessing subjective psychological well-being based on respondent ratings of cheerfulness, calmness, feelings of vigor, feelings of being well rested after sleep, and personal interest. Responses are provided on a 6-point scale: 0 ("at no time") to 5 ("all of the time") according to the proportion of time over the preceding 2 weeks that applied to each attribute. Scores range from 0-25; higher scores reflect better well-being.
Change in Breslau Post Traumatic Stress Disorder (PTSD) Scores | Day 1, Day 180
  The Breslau Post Traumatic Stress Disorder screen is a 7-symptom measure assessing presence of PTSD in accordance with Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) and World Health Organization guidelines. Responses are provided on a 2-point scale: 1 ("Yes") or 0 ("No") in response to 7 questions. Scores of 4 or more indicate a likelihood of PTSD.
Change in Perceived Stress Scale (PSS-4) Scores | Day 1, Day 180
  The Perceived Stress Scale is a 4-item measure, self-report scale that generates a global stress score based on general questions rather than specific experiences. Response are provided on a 5-point scale: 0 ("Never") to 4 ("very often") according to the proportion of time over the preceding month that applied to each attribute. Scores range from 0-16. Scores of 0-7 indicate low to moderate stress; scores of 8-16 indicate moderate to high stress level.
Change in Utrecht Work Engagement Scale (UWES) Scores | Day 1, Day 180
  The UWES is a 3-item measure assessing engagement in an individual's work based on respondent ratings of vigor, dedication, and absorption. Responses are provided on a 7-point scale: 0 ("never") to 6 ("always, every day") and averaged. Scores range from 0-6; scores within 0-4 indicate low engagement and satisfaction in the workplace.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9-36 months
Access Criteria: Approval from an investigator's IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Kennedy S, Carmack S, Li L, Lin FC, Hatch JE, Chan K, Tolleson-Rinehart S, Noah TL. Coaching Pediatricians for Wellbeing: A Pilot Feasibility and Acceptability Study. Acad Pediatr. 2025 Mar;25(2):102586. doi: 10.1016/j.acap.2024.09.010. Epub 2024 Oct 1. PMID 39362630